CLINICAL TRIAL: NCT04457674
Title: Targeting Sleep Homeostasis to Improve Alcohol Use Disorder Treatment Outcomes
Brief Title: Targeting Sleep Homeostasis to Improve Alcohol Use Disorder Treatment Outcomes (M-STAR Study)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, J. Todd Arnedt, Associate Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00173631; R01AA028158 (NIH)
Record Dates: First submitted 2020-06-29; First posted 2020-07-07 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-07

CONDITIONS: Insomnia; Alcohol Use Disorder
Keywords: Cognitive Behavioral Therapy; Sleep Hygiene
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Alcoholism; Sleep Hygiene | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy for insomnia (CBTi) (Other): CBTi is a non-medication therapy that includes cognitive and behavioral treatment components.
  Interventions: Behavioral: Cognitive Behavioral Therapy for insomnia (CBTi)
- Sleep Hygiene Education (SHE) (Other): SHE is a non-medication therapy that focuses on identifying and changing several behavioral and environmental factors that can interfere with sleep.
  Interventions: Behavioral: Sleep Hygiene Education (SHE)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for insomnia (CBTi) — CBTi consists of six weekly sessions of individual therapy with a trained therapist, delivered via telemedicine.
  Arms: Cognitive Behavioral Therapy for insomnia (CBTi)
Behavioral: Sleep Hygiene Education (SHE) — SHE participants receive six weekly sessions of individual therapy with a trained therapist, delivered via telemedicine.
  Arms: Sleep Hygiene Education (SHE)

SUMMARY:
Insomnia is common in people who are in treatment for alcohol use disorder. It can impact both sleep quality and daytime functioning, as well as make it harder to treat the underlying alcohol use disorder. This study is looking at two types of therapy to help manage insomnia specifically for people also in treatment for alcohol use disorder.

ELIGIBILITY:
Inclusion Criteria:

* Meet probable Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria for Alcohol Use Disorder with ≤12 months of abstinence
* Planned enrollment into an abstinence-based treatment program
* Meet probable DSM-5 criteria for chronic insomnia
* Access to a video chat-capable device and reliable Wi-Fi network

Exclusion Criteria:

* Diagnosis of, or high suspicion for, sleep disorders other than insomnia
* Meet probable DSM-5 criteria for bipolar disorder, psychotic disorder, or post-traumatic stress disorder (PTSD)
* Terminal or progressive physical illness (e.g., cancer), neurological degenerative disease (e.g., dementia), or presence of an unstable medical condition that is the specific cause of insomnia
* Self-reported pregnancy or intention to become pregnant during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Score from the insomnia severity index (ISI) | Immediately post treatment
  The ISI is a 7-item self-report assessment of the nature, severity and impact of insomnia. Scores range from 0-28 with higher scores suggesting more clinically significant insomnia.
Percent days abstinent from alcohol as documented in the timeline follow-back (TLFB) | Immediately post treatment
  The Alcohol TLFB is an interviewer-based drinking assessment method to estimate drinking behaviors, including both frequency and quantity of consumption.

SECONDARY OUTCOMES:
Score from Multidimensional Fatigue Inventory (MFI), General Fatigue sub-scale | Immediately post treatment
  The MFI is a 20-item assessment that provides an overall fatigue score (20-100) in addition to 5 separate dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. Sub-scale scores range from 4-20 with higher scores indicating higher levels of fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: J Todd Arnedt, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared through the National Institute of Mental Health (NIMH) Data Archive. Only information relevant to the research project will be shared, which may include demographic information such as gender and age, responses to surveys and results found from the research project. Participants identifying data will not be shared in any way and information related to participants will be given a different random identifier known as a Global Unique Identifier or GUID. This number will not coincide with any identifier for data stored on University of Michigan study databases.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available following data collection and for 1-2 years following the end of the study grant.
Access Criteria: Data shared via the NIMH database is accessible by those associated with NIH institutions who have also signed data sharing agreements.

DOCUMENTS (1):
  • Informed Consent Form (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/74/NCT04457674/ICF_000.pdf